CLINICAL TRIAL: NCT01927536
Title: Evaluating Color Perception Under LED Red/Green and Green Dominant Light
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0387
Record Dates: First submitted 2013-08-02; First posted 2013-08-22 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Color Blindness, Acquired
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Night Vision: White LED Flashlight, Red/Green Green Dominant LED Flashlight
  Interventions: Device: White LED Flashlight; Device: Red/Green Green Dominant LED Flashlight

INTERVENTIONS:
Device: White LED Flashlight — white light setting
  Other Names: Tomahawk serial number TMC12420
Device: Red/Green Green Dominant LED Flashlight — Green LED light dominant setting
  Other Names: Tomahawk serial number TMC12420, green dominant setting

SUMMARY:
The investigators are testing a Light-emitting Diode (LED) flashlight from First-Light™ USA called the Tomahawk MC Tactical Light to determine the range of colors people are able to see with these flashlights at night. The flashlight has been designed to reduce visibility of the user and uses a combination of green and red LED lamps to achieve this. In this study investigators wish to determine how well a subject can differentiate colors at night in a quantifiable manner. Investigators will use the Farnsworth Munsell 100 hue test which requires the user to put shades of red, green, blue and yellow into progressive color order which is scored according to the manufactures specifications.

ELIGIBILITY:
Inclusion Criteria:

* normal vision
* 18-65 years

Exclusion Criteria:

* blindness
* colorblind
* pregnant women
* prisoners
* decisionally challenged

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal color vision status
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Normal Color vision | 1 hr
  The Farnsworth Munsell 100 Hue Test is used to determine normal color vision and vision using the red green Tomahawk LED flashlight.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Petrash, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Dept of Opthalmology, Aurora, Colorado, United States